CLINICAL TRIAL: NCT05772169
Title: Study of Hypercortisolism in Patients With Difficult to Control Type 2 Diabetes Despite Receiving Standard-of-Care Therapies: Prevalence and Treatment With Korlym® (Mifepristone) (CATALYST)
Brief Title: Study to Determine the Prevalence of Hypercortisolism in Patients With Type 2 Diabetes and Treatment With Korlym® (Mifepristone) (CATALYST)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-1073-310
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Hypercortisolism; Diabetes Mellitus, Type 2
Keywords: Hypercortisolism; Diabetes Mellitus, Type 2 Uncontrolled
MeSH Terms: conditions — Cushing Syndrome; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mifepristone 300 mg (Experimental): Randomized to receive 300 mg mifepristone, titrated to 600 mg mifepristone after 4 weeks with an opportunity to increase to 900 mg mifepristone at week 8 or 12
  Interventions: Drug: Mifepristone 300 MG [Korlym]
- Placebo (Placebo Comparator): Patients who meet the entry criteria for the Study C-1073-310 will be randomized to receive placebo for 24 weeks
  Interventions: Drug: Placebo for mifepristone

INTERVENTIONS:
Drug: Mifepristone 300 MG [Korlym] — Mifepristone tablets for once daily oral dosing
  Arms: Mifepristone 300 mg
Drug: Placebo for mifepristone — Placebo tablets for once daily oral dosing
  Arms: Placebo

SUMMARY:
This is a Phase 4 study with 2 parts: Part 1 (Prevalence Phase) is non-interventional and will assess the prevalence of hypercortisolism in a population with difficult to control type 2 diabetes (T2D) (hemoglobin A1c ≥7.5%) despite receiving standard-of-care therapies. Part 2 (Treatment Phase) is a randomized, prospective, placebo-controlled, double-blind multi-center trial that will assess the safety and efficacy of mifepristone treatment in patients with hypercortisolism who have difficult to control T2D despite receiving standard of care therapies.

DETAILED DESCRIPTION:
This is a Phase 4 study with 2 parts at approximately 30 sites in the United States (US).

Part 1 (Prevalence Phase) is non-interventional and will assess the prevalence of hypercortisolism in a population with difficult to control T2D (HbA1c ≥7.5%) despite receiving standard-of-care therapies.

Patients from Part 1 Prevalence Phase who meet eligibility requirements can then enroll in Part 2 and will be randomized 2:1 to receive mifepristone or placebo once daily with food. Randomization will be stratified by presence of adenoma (yes/no).

Part 2 (Treatment Phase) is a randomized, prospective, placebo-controlled, double-blind multi-center trial that will assess the safety and efficacy of mifepristone treatment in patients with hypercortisolism who have difficult to control T2D despite receiving standard of care therapies.

ELIGIBILITY:
For Part 1:

Inclusion Criteria:

Has difficult to control T2D (HbA1c ≥7.5% and ≤11.5%) based on HbA1c performed at screening.

AND Taking 3 or more anti-hyperglycemic drugs. OR Taking insulin and other anti-hyperglycemic drugs. OR Taking 2 or more anti-hyperglycemic drugs AND a.) the presence of 1 or more micro-vascular or macro-vascular complication (retinopathy, diabetic nephropathy and chronic kidney disease, diabetic neuropathy, atherosclerotic heart disease with diabetes); AND/OR b.) concomitant hypertension requiring 2 or more anti-hypertension medications.

• Women on oral contraceptive pills (OCPs) may be screened but must be willing and able to stop OCPs for at least 3 weeks prior to the dexamethasone suppression test.

Exclusion Criteria:

* Has type 1 diabetes mellitus.
* New-onset diabetes less than 1 year.
* Systemic glucocorticoid medications exposure (excluding inhalers or topical) within 3 months of screening.
* Is pregnant or lactating. For women of childbearing potential, have a positive pregnancy test before dexamethasone administration. A woman of childbearing potential includes all women <50 years old, women whose surgical sterilization was performed <6 months ago, and women who have had a menstrual period in the last 12 months.
* On hemodialysis or has end-stage renal disease.
* Has severe untreated sleep apnea as judged by the Investigator.
* Has excessive alcohol consumption (>14 units/week for male, >7 units/week for female) as judged by the Investigator.
* Has severe psychiatric illness by history (such as schizophrenia or dementia) as judged by the Investigator.
* Has severe medical or surgical illness as judged by the Investigator.
* Is a night shift worker, i.e., is awake from approximately 11 PM to 7 AM.
* Has taken any investigational drug within 4 weeks prior to screening, or within less than 5 times the drug's half-life, whichever is longer.
* Has had the diagnosis of Cushing syndrome or has used or plans to use any of the following treatments for Cushing syndrome:

  - Mifepristone, metyrapone, osilodrostat, ketoconazole, fluconazole, aminoglutethimide, etomidate, octreotide, larazotide, pasireotide, long-acting octreotide or pasireotide.
* Has a history of hypersensitivity or severe reaction to dexamethasone

For Part 2:

Inclusion Criteria:

* Has completed Part 1 of the study with post-DST cortisol level of >1.8 μg/dL and dexamethasone level ≥140 ng/dL
* Will have no change in, or initiation of, diabetes medications within 4 weeks prior to first study drug dose

Exclusion Criteria:

* Has any change in status of exclusion criteria from Part 1
* Requires inhaled glucocorticoid use and may require systemic glucocorticoids if their condition deteriorates during study
* Has severe, poorly controlled hypertension at screening (defined as mean systolic BP >160 mmHg or mean diastolic BP >100 mmHg); must be able to correct to a BP of <160/100 mmHg before first dose of study drug
* Has refractory hypokalemia; must be able to correct to potassium level of ≥4.0 mEq/L before first dose of study drug
* Has poorly controlled hyperthyroidism/hypothyroidism before first dose of study drug (confirmed by TSH or free thyroxine)
* Has plans for adrenalectomy or adrenal nodulectomy
* Has renal insufficiency (eGFR <30 mL/min/1.73m2)
* Has liver test results >3x ULN (ALT or AST) or bilirubin >1.5x ULN
* Takes drugs metabolized by CYP3A and CYP3A substrates with narrow therapeutic ranges
* Receiving systemic corticosteroids that cannot be discontinued
* Uses hormonal contraceptives
* Has a history of unexplained vaginal bleeding, endometrial hyperplasia with atypia, or endometrial carcinoma
* Is pregnant or lactating
* Has a known hypersensitivity to mifepristone or any of the product components

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1113 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Part 1 Prevalence Phase: Prevalence of Hypercortisolism | Screening
  Prevalence (percentage) of patients with hypercortisolism defined by dexamethasone suppression test (DST) >1.8 μg/dL with dexamethasone level ≥140 ng/dL in patients with difficult to control T2D, defined as HbA1c ≥7.5%. despite receiving standard-of-care therapies.
Part 2 Treatment Phase: Effect of Treatment on Hypercortisolism with Abnormal Adrenal CT Scan | Baseline Day 1 to week 24
  Change in HbA1c from baseline (at randomization) to 24 weeks in patients with hypercortisolism and abnormal adrenal CT scan who have difficult to control T2D despite receiving standard of care therapies, treated with mifepristone versus placebo.
Part 2 Treatment Phase: Effect of Treatment on Hypercortisolism without Abnormal Adrenal CT Scan | Baseline Day 1 to week 24
  Change in HbA1c from baseline (at randomization) to 24 weeks in patients with hypercortisolism and normal adrenal CT scan who have difficult to control T2D despite receiving standard of care therapies, treated with mifepristone versus placebo.

SECONDARY OUTCOMES:
Part 1 Prevalence Phase: Origin of Hypercortisolism | Screening
  Percentage of patients with/without abnormal adrenal CT scan.
Part 1 Prevalence Phase: Patient Characteristics | Screening
  Clinical and/or laboratory characteristics of patients with hypercortisolism and of patients with hypercortisolism with/without abnormal adrenal CT scan.
Part 2 Treatment Phase: Effect of Treatment | Baseline Day 1 to week 24
  Change in anti-diabetes medication from baseline (at randomization) to 24 weeks in patients with hypercortisolism with/without abnormal adrenal CT scan who have difficult to control T2D despite receiving standard-of-care therapies, treated with mifepristone versus placebo.
Part 2 Treatment Phase: Effect of Treatment | Baseline Day 1 to week 24
  Change from baseline (at randomization) to 24 weeks in body weight, body mass index, waist circumference, other glycemic metrics, blood pressure, quality of life, antihypertensive medications, etc. in patients with hypercortisolism with/without abnormal adrenal CT scan treated with mifepristone versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Einhorn, MD, Study Director — Corcept Therapeutics
Locations (36):
- United States (36):
  - Site 407, Escondido, California
  - Site 379, Gardena, California
  - Site 378, Huntington Park, California
  - Site 406, La Jolla, California
  - Site 373, Los Angeles, California
  - Site 387, Tarzana, California
  - Site 375, Torrance, California
  - Site 444, Edgewater, Florida
  - Site 015, Fort Lauderdale, Florida
  - Site 009, Atlanta, Georgia
  - Site 097, Atlanta, Georgia
  - Site 046, Covington, Kentucky
  - Site 061, Metairie, Louisiana
  - Site 377, New Orleans, Louisiana
  - Site 205, New Orleans, Louisiana
  - Site 410, Baltimore, Maryland
  - Site 394, Hyattsville, Maryland
  - Site 067, Boston, Massachusetts
  - Site 074, Ann Arbor, Michigan
  - Site 371, Las Vegas, Nevada
  - Site 070, Albany, New York
  - Site 411, Smithtown, New York
  - Site 181, Chapel Hill, North Carolina
  - Site 059, Wilmington, North Carolina
  - Site 436, Cincinnati, Ohio
  - Site 042, Cleveland, Ohio
  - Site 077, Columbus, Ohio
  - Site 195, Columbus, Ohio
  - Site 435, Grants Pass, Oregon
  - Site 049, Portland, Oregon
  - Site 456, Cedar Park, Texas
  - Site 370, Dallas, Texas
  - Site 408, Lufkin, Texas
  - Site 054, San Antonio, Texas
  - Site 369, San Antonio, Texas
  - Site 405, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Upon study completion, results will be presented at relevant scientific congresses and published in a peer-reviewed journal.

REFERENCES:
- [Derived] DeFronzo RA, Auchus RJ, Bancos I, Blonde L, Busch RS, Buse JB, Findling JW, Fonseca VA, Frias JP, Hamidi O, Handelsman Y, Pratley RE, Rosenstock J, Tudor IC, Moraitis AG, Einhorn D. Study protocol for a prospective, multicentre study of hypercortisolism in patients with difficult-to-control type 2 diabetes (CATALYST): prevalence and treatment with mifepristone. BMJ Open. 2024 Jul 16;14(7):e081121. doi: 10.1136/bmjopen-2023-081121. PMID 39013654